CLINICAL TRIAL: NCT01254838
Title: Novel Peptide Vaccination for Patients With Advanced Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Iwate Medical University (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Departmet of Urology, Iwate Medical University
Other Study IDs: IMU-H20-30-P1
Record Dates: First submitted 2010-12-02; First posted 2010-12-07 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2008-11

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: HLA-A02 restricted HIG2

SUMMARY:
The purpose of this study is to evaluate the safety and CTL reaction of novel peptide vaccination for advanced renal cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS advanced renal cell carcinoma which already showed resistance to standard treatments

PATIENTS CHARACTERISTICS

1. Patients who showed resistance to hormonal therapy and chemotherapy
2. Histological diagnosis is adenocarcinoma
3. HLA-A*0201/0206
4. ECOG performance status of 0 to 2
5. Age ≥ 20 years, ≤80 years
6. WBC≥ 2,000/mm³, ≤12000/mm³ hemoglobin≥ 8.0g/dl Platelet count ≥ 70000/mm³ AST, ALT ≤100 IU/l Total bilirubin ≤ 1.5 mg/dl Creatinine ≤ 1.0 mg/dl PaO2≥ 70mmHg
7. life expectancy ≥ 3months
8. Able and willing to give valid written informed consent

Exclusion Criteria:

1. Pregnancy (women of childbearing potential: Refusal or inability to use effective means of contraception)
2. Breastfeeding
3. Patients willing to childbearing ( Refusal or inability to use effective means of contraception)
4. Serious infections requiring antibiotics
5. Concomitant treatment with steroids or immunosuppressing agent
6. Other malignancy difficult to control.
7. Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2008-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2 years
  hematological and non-hematological adverse event

SECONDARY OUTCOMES:
CTL reaction | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Tomoaki Fujioka, Study Chair — Department of Urology, Iwate Medical University